CLINICAL TRIAL: NCT01027416
Title: Pilot Study to Analyze a Novel Mechanism Underlying Response to Tamoxifen Therapy in Breast Cancer Patients
Brief Title: Analyzing a New Mechanism in Response to Tamoxifen Therapy in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RPCI I 110907; R21CA137635-01A1 (NIH); NCT01658566 (obsolete NCT alias)
Record Dates: First submitted 2009-12-04; First posted 2009-12-08 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer
Keywords: ER positive; Tamoxifen
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Intervention (No Intervention)
- Tamoxifen (Active Comparator): Tamoxifen 20 mg orally 1x/day for 4 weeks
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Tamoxifen — Drug: Tamoxifen 20 mg orally 1x/day for 4 weeks
  Arms: Tamoxifen

SUMMARY:
This study will help to understand the interaction between estrogen receptor-alpha (ER alpha) and tumor suppressor protein p53 as well as impact on patient tumor gene expression in response to the hormonal therapy Tamoxifen. This information may eventually help select the appropriate therapy for future patients with similar cancer.

DETAILED DESCRIPTION:
Women with abnormal mammogram or suspicious masses will undergo diagnostic core biopsies which will be analyzed for ER/PR and HER2Neu expression. For patients that are ER positive, p53 staining will be done.

Women presenting tumors with an Allred score of 3 or greater status will be approached to participate.

Women will be randomized to either standard of care surgical therapy or a 4 week intervention of Tamoxifen 20mg daily for 4 weeks prior to surgery. During the intervention, blood draws will be done to measure levels of tamoxifen metabolites in the blood and test for polymorphisms that may decrease levels of active metabolites.

Women will undergo two blood draws for PK/PD and one for pharmacogenomics. Tissue microarray (TMA) will be generated from resected tumors for immunohistochemistry (IHC) and proximity ligation assay (PLA) for measuring ER alpha-p53 interaction.

Tumor tissue will be used for analyzing tamoxifen metabolites and estradiol levels. RNA and proteins from the tumors will be used for analyzing gene expression.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must consent to be in the study and must have signed an approved consent form conforming to institutional guidelines
2. The patient must be 18 years or older.
3. Core biopsy should definitively demonstrate invasive carcinoma.
4. Invasive carcinoma should be ER-apha receptor positive
5. The tumor should be approximately at least 1 cm, to account for variability in imaging and imaging occult disease (physical exam, mammography, ultrasound). We recognize that from time to time because of this variation, there might not be enough tissue available for analysis after surgical excision but this will allow the greatest opportunity to capture as many eligible patients as possible.
6. Patients in whom surgical excision of the tumor is part of standard of care management
7. ECOG score of 0 or 1
8. Negative serum or urine beta-hCG pregnancy test at screening for patients of child-bearing potential (this is routinely done if the patient is premenopausal and having surgery)
9. Consent to participate in DBBR (RPCI only)

Exclusion Criteria:

1. Male patients are not eligible for this study
2. Female patients with inoperable tumors or women with stage 4 disease diagnosed on CT, PET, PET/CT or bone scan.
3. Patients with diagnosis by FNA cytology only
4. Pregnant or lactating women
5. Prior therapy for breast cancer, including irradiation, chemo- immuno- and/or hormonal therapy
6. Patients receiving any hormonal therapy, e.g. ovarian hormonal replacement therapy, infertility medications etc., are not eligible
7. Nonmalignant systemic disease (cardiovascular, renal, hepatic, etc.) that would preclude the patient from being subjected to surgical excision
8. Psychiatric or addictive disorders that would preclude obtaining informed consent
9. Patients known or suspected to have hypercoagulable syndrome or with history of venous or arterial thrombosis, stroke, TIA, or pulmonary embolism
10. Women with non-invasive disease or microinvasion are not eligible.
11. Women undergoing neoadjuvant chemotherapy are not eligible
12. women currently on tamoxifen and raloxifene for prevention are not eligible
13. Patients shall not receive any herbal/alternative therapies such as flaxseed or soy products or black cohosh.
14. Patients with a known mutation in p53 (Li Fraumeni Syndrome)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2009-12-14 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gokul Das, PhD, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - University of Chicago, Chicago, Illinois
  - Roswell Park Cancer Institute, Buffalo, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- No Intervention: No Intervention: Standard of care
Period: Overall Study
Arm/Group | No Intervention | Tamoxifen
Started | 31 | 28
Completed | 30 | 23
Not Completed | 1 | 5
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 1 | 4

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | No Intervention | Tamoxifen | Total
Number analyzed (Participants) | 31 | 28 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 19 | 44
  >=65 years | 6 | 9 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (11.1) | 58.5 (12.4) | 57.0 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 28 | 59
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 27 | 23 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Positive Proximity Ligation Assays of All Tumor Protein p53-wild Type Breast Tumors in Participants by Treatment Arm
Description: Status of estrogen receptor alpha (ERά) and tumor protein (p53) interaction in p53-wild type breast tumors in untreated patients verses patients treated with tamoxifen. Mean percent positive polylactide (PLA) of all p53-wild type breast tumors in participants by treatment arm
Time Frame: 2 years
Population: All patients with p53-wild type breast tumors
Measure: Mean (Standard Deviation); unit: percentage of positive PLA
Arm/Group | No Intervention | Tamoxifen
Number analyzed (Participants) | 23 | 12
percentage of positive PLA | 27.0 (34.4) | 4.4 (4.4)

2. Secondary Outcome: Total Number of Over-expressed Genes, Across All Participants With Tumor Protein p53-wild Type Breast Tumors That Had RNA Samples Available.
Description: Total number of over-expressed genes, across all participants with tumor protein p53-wild type breast tumors that had ribonucleic acid (RNA) samples available.
Time Frame: 2 years
Population: All patients with p53-wild type breast tumors that had RNA samples available
Measure: Number; unit: genes
Arm/Group | No Intervention | Tamoxifen
Number analyzed (Participants) | 20 | 15
genes | 196 | 256

ADVERSE EVENTS:
Arm/Group | No Intervention | Tamoxifen
Serious Adverse Events (participants affected / at risk) | 1/31 | 0/28
Other Adverse Events (participants affected / at risk) | 0/31 | 19/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Intervention (N=31) | Tamoxifen (N=28)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Intervention (N=31) | Tamoxifen (N=28)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 4 (6)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 5 (5)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 5 (7)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 6 (8)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (5)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 7 (10)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 5 (5)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (9)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 6 (8)
Fatigue (General disorders) | 0 (0) | 3 (4)
Irritability (General disorders) | 0 (0) | 8 (10)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 4 (5)
Sensation of pressure (General disorders) | 0 (0) | 1 (1)
Surgical failure (General disorders) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 1 (3)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 5 (7)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Disturbance in attention (Nervous system disorders) | 0 (0) | 6 (6)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 9 (14)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 7 (8)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Neurological symptom (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Bladder discomfort (Renal and urinary disorders) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 2 (3)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 3 (4)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 9 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Hot flush (Vascular disorders) | 0 (0) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-23): https://cdn.clinicaltrials.gov/large-docs/16/NCT01027416/Prot_SAP_000.pdf